CLINICAL TRIAL: NCT07126470
Title: Effect of Capsular Tension Ring Implantation on Postoperative IOL Position in Retinitis Pigmentosa Patients With Cataract: a Single-center, Randomized, Self-controlled Study
Brief Title: Impact of Capsular Tension Ring on Intraocular Lens Position in Retinitis Pigmentosa Cataract Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025KYPJ066
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cataract; Retinitis Pigmentosa (RP)
MeSH Terms: conditions — Cataract; Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: This is an intraindividual comparative study. Each participant receives bilateral cataract surgery, with one eye randomly assigned to CTR implantation and the other eye without CTR.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group: IOL Plus CTR implantation (Experimental): Patients will undergo phacoemulsification combined with IOL and CTR implantation
  Interventions: Procedure: CTR implantation
- Control Group: IOL implantation Only (No Intervention): Patients will undergo phacoemulsification combined with IOL implantation. All patients undergo uneventful phacoemulsification by a 2.2 mm temporal transparent corneal incision using Centurion Vision System (Alcon Laboratories, Fort Worth, TX, USA). After the nucleus and cortex are removed, IOL (J&J Tecnis DCB00) is implanted in the capsular bag.

INTERVENTIONS:
Procedure: CTR implantation — Device: CTR (275001G, OPHTEC BV, Netherlands) All patients undergo uneventful phacoemulsification by a 2.2 mm temporal transparent corneal incision using Centurion Vision System (Alcon Laboratories, Fort Worth, TX, USA). After the nucleus and cortex are removed, a capsular tension ring is implanted in the capsular bag and then IOL (J&J Tecnis DCB00) is implanted.
  Arms: Treatment Group: IOL Plus CTR implantation

SUMMARY:
This is a self-controlled randomized clinical trial to investigate the effect of capsular tension ring (CTR) implantation on intraocular lens (IOL) position in cataract patients with retinitis pigmentosa(RP). Each patient will receive CTR implantation in one eye, with the fellow eye serving as control. Postoperative outcomes, including visual acuity, IOL position, and postoperative complications will be compared between eyes.

DETAILED DESCRIPTION:
Patients with retinitis pigmentosa (RP) have a higher risk of developing cataracts, often accompanied by abnormalities such as zonular laxity and vitreous liquefaction, which increases the risk of intraocular lens (IOL) tilt, decentration, and capsular contraction after surgery. The capsular tension ring (CTR) can support the zonules and maintain the stability of the capsular bag, but its effect in RP patients remains controversial.

In this self-controlled clinical trial, we are going to recruit 88 RP patients scheduled for bilateral cataract surgery. Both eyes receive a monofocal DCB00 IOL, while only on eye receives an additional CTR. Follow up visits take place 1 week, 1 month, 3 months, 6 months, and 1 year postoperatively. At the follow up visits, IOL decentration and tilt (determined by anterior segment SS-OCT Casia 2), visual acuity, and postoperative complications will be compared intraindividually at different timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Clinical diagnosis of retinitis pigmentosa (RP).
* Bilateral cataract meeting the indications for IOL implantation.
* Willingness to participate in the study and provision of signed informed consent.

Exclusion Criteria:

* History of intraocular surgery.
* Severe zonular weakness (e.g., zonular dialysis >90°, lens subluxation/dislocation)
* Other ocular comorbidity: such as pseudoexfoliation syndrome, ocular trauma, corneal dystrophies, uveitis, etc.
* Severe systemic diseases: such as severe hypertension, diabetes, heart disease, Alzheimer's, Parkinson, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
IOL dencentration | 3 months after surgery
  Measured by anterior segment OCT (CASIA2)

SECONDARY OUTCOMES:
IOL dencentration | Baseline (before surgery), 1 week, 1 month, 6 months, 1 year after surgery
  Measured by anterior segment OCT (CASIA2)
IOL tilt | Baseline (before surgery), 1 week, 1 month, 3 months, 6 months, 1 year after surgery
  Measured by anterior segment OCT (CASIA2)
BCVA | Baseline (before surgery), 1 week, 1 month, 3 months, 6 months, 1 year after surgery
  BCVA is evaluated with ETDRS visual acuity chart.
Postoperative complications | 1 week, 1 month, 3 months, 6 months, 1 year after surgery
  Postoperative complications such as posterior capsular opacification, anterior capsule contraction, cystoid macular edema are examined by slit lamp photograph and other devices if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Tan, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No